CLINICAL TRIAL: NCT05752942
Title: Precision-Based Approach to Matching Evidence-Based Interventions to Individual Needs of Students With Externalizing Behaviors: A Double-Masked Randomized Controlled Trial
Brief Title: Precision-Based Approach to Matching Evidence-Based Interventions to Students With Externalizing Behaviors
Acronym: SIMSRCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Collaborators: University of Minnesota (Other)
Responsible Party: Principal Investigator, Yanchen Zhang, Assistant Professor, University of Iowa
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SIMS001
Record Dates: First submitted 2023-02-21; First posted 2023-03-03 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: Problem;Behaviour;Child

STUDY DESIGN:
Intervention Model Description: single-level two-arm randomized waitlist-controlled trial
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment: Student Intervention Matching System (Experimental): In the treatment condition, the students received a performance-based interventions matched to their individual needs and characteristics based on Student Intervention Matching System (SIMS).
  Interventions: Behavioral: Student Intervention Matching System (SIMS)
- Active control: group-based social skills training (Active Comparator): In the control condition, students received an unconditionally mismatched acquisition-based EBI (group-based social skills training).
  Interventions: Behavioral: group-based social skills training

INTERVENTIONS:
Behavioral: Student Intervention Matching System (SIMS) — The Student Intervention Matching System (SIMS) is a pre-intervention matching assessment following the behavioral consultation model. The SIMS entails three steps to sequentially assess and then match students' individual characteristics to precise acquisition- or performance-based interventions. The 1st step corresponds to the "problem identification" stage in behavioral consultation. The 2nd step corresponds to the "problem analysis" stage of behavioral consultation.The 3rd step of SIMS corresponds to the "implementation planning" and "evaluation" stages of behavioral consultation.
  Arms: Treatment: Student Intervention Matching System
Behavioral: group-based social skills training — In the control condition, students received an unconditionally mismatched acquisition-based intervention (group-based social skills training). We selected group-based social skills training for four reasons: (a) participating schools had already been delivering it as their treatment-as-usual, (b) it is a common intervention in US schools, (c) it is only effective for students with acquisition needs, and (d) it represents a counterfactual contrast to the treatment condition because externalizing behaviors driven by performance needs will be reduced more by performance-based interventions than acquisition-based ones.
  Arms: Active control: group-based social skills training

SUMMARY:
Although prevalent across schools in the US, the "One-Size-Fits-All" (OSFA) approach to selecting evidence-based interventions (EBIs) for student externalizing behaviors often yields lackluster outcomes, due to the mismatch between the EBI and students' heterogeneous needs. Emerging literature highlighted the promise of the precision approach to intervention (e.g., Student Intervention Matching System; SIMS), whereas EBIs were selected based on the match between a student's individual needs and the active components of EBIs. This pilot study tested the efficacy, feasibility, and acceptability of SIMS to match EBIs to students with externalizing behaviors. The investigators ran a double-masked randomized waitlist-controlled trial in a diverse urban district. Students at risk for externalizing behaviors were recruited and randomly assigned to the treatment (EBIs matched via SIMS) or control condition (mismatched social-skill training). Students received EBIs based on assigned condition for 10 weeks. Students' externalizing behaviors were assessed via a multi-method approach at baseline and 10-week posttest. Teachers rated the feasibility and acceptability of SIMS at 10-week posttest. The investigators used cluster-adjusted ANCOVAs to compare efficacy of matched EBIs via SIMS against that of the mismatched social skill training in reducing student externalizing behaviors.

ELIGIBILITY:
Inclusion Criteria:

* with a moderate risk for externalizing behavioral problems, which was indicated by a score between 4 and 8 on the Student Risk Screening Scale-Externalizing.
* receiving the majority of services in general education settings
* in 3rd, 4th, or 5th grade level.

Exclusion Criteria:

* severe risk for externalizing problems, which was indicated by a score exceeding 8 on the Student Risk Screening Scale-Externalizing. The students at severe risk will be referred to the school counselor for appropriate service.

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 51 (Actual)
Dates: Start 2018-08-25 (Actual); Primary Completion 2018-11-10 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Change in the frequency of students' externalizing behaviors from baseline to 10-week follow-up | Start of the study (baseline) and End of the study (10-week posttest)
  The Direct Behavior Rating- Multi-Item Scale (DBR-MIS) is a pragmatic and low-inference assessment of an operationally defined problem behavior on a specific dimension (frequency, intensity, or duration of externalizing behaviors; Christ et al., 2009). The educators complete the DBR-MIS based on their observations of the target student in the setting where the problem behavior usually occurs for a pre-specified period. The DBR-MIS contains three items corresponding to disruptive behaviors, aggressive behavior, and noncompliance, which were summed into a total score of externalizing behaviors. Each item was rated on a 10-point Likert scale ranging from "0%; Never" to "50%; Sometimes" to "100%; Always".
Change in the severity of students' externalizing behaviors from baseline to 10-week follow-up | Start of the study (baseline), and End of the study (10-week posttest)
  The Social Skills Improvement System-Rating Scale (SSIS-RS; Elliott et al., 2008) is a brief and intervention-oriented assessment of students' needs in social skills and problem behaviors. Given the scope of this study, only the "externalizing behavior subscale" were used. Each item was rated on a 3-point Likert scale (0= Never, 1= Seldom, 2 = Often, and 3= Almost Always) based on the frequency of a student's externalizing behavior. High scores indicate more frequent externalizing behaviors.

SECONDARY OUTCOMES:
Feasibility and Acceptability | End of the study (10-week posttest)
  The school teams and designated implementers of matched EBIs rated the feasibility and acceptability of the EBIs matched via SIMS. Given the scope of this study, we used two subscales, Feasibility (7-item) and Acceptability (9-item), from the Usage Rating Profile-Intervention Revised (URP-IR; Chafouleas et al., 2011). All items were rated on a 6-point Likert scale ranging from 1 "strongly disagree" to 6 "strongly agree".
Intervention Fidelity | End of the study (10-week posttest)
  The designated implementers of matched EBIs (e.g., teachers, paraprofessionals, or behavioral specialists) used EBI-specific checklists to assess their intervention fidelity. Given the scope of this study and the common practice in school-based intervention research, we used implementers' adherence to the EBI protocols as the primary indicator of intervention fidelity. Fidelity checklists were developed by (a) operationalizing the core components of an EBI, and (b) having implementers to self-report how many core components they delivered as intended for the target student during a specific period.

CONTACTS AND LOCATIONS:
Overall Officials: Clayton Cook, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota-Twin Cities, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified datasets generated and analyzed during the current study are available upon request to the principle investigator.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: From February 1st, 2023 with no ending date.
Access Criteria: Public upon request to the principle investigator

REFERENCES:
- [Background] Chafouleas SM. Direct Behavior Rating: A review of the issues and research in its development. Education and Treatment of Children. 2011;34(4):575-91.
- [Background] Elliott SN, Gresham FM, Frank JL, Beddow III PA. Intervention validity of social behavior rating scales: Features of assessments that link results to treatment plans. Assessment for effective intervention. 2008 Dec;34(1):15-24.
- [Background] Christ TJ, Riley-Tillman TC, Chafouleas SM. Foundation for the development and use of Direct Behavior Rating (DBR) to assess and evaluate student behavior. Assessment for Effective Intervention. 2009 Sep;34(4):201-13.